CLINICAL TRIAL: NCT05237583
Title: Does a Multimodal Prehabilitation Program Improve Markers of Frailty in Patients With Cirrhosis Undergoing Liver Transplantation? A Feasibility Trial
Brief Title: Prehabilitation for Patients Awaiting Liver Transplantation
Acronym: Prehab preLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Donation and Transplantation Research Program (Unknown); Canadian Association for the Study of the Liver (Unknown)
Responsible Party: Principal Investigator, Amine Benmassaoud, Study Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-7646
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cirrhosis, Liver; Liver Transplantation; Frailty
Keywords: Prehabilitation; Nutrition; Quality of life; Exercise; Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Frailty; Motor Activity; Fibrosis | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): Multimodal prehabilitation program
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — All participants will be offered a multimodal prehabilitation program. This program will include an individualized and supervised aerobic and resistance exercise training program, nutritional optimization, and psychological support. The program will last 6 months or until liver transplantation, whichever comes first.

SUMMARY:
This study will assess the feasibility, safety and effectiveness of a structured prehabilitation program combining exercise training, nutritional optimization and psychological support for patients with cirrhosis awaiting liver transplantation.

DETAILED DESCRIPTION:
Due to their chronic liver disease, patients with cirrhosis awaiting liver transplantation develop low muscle mass, poor nutritional status and decreased reserves putting them at high risk of postoperative complications, prolonged hospital stay, and failed discharge home after liver transplantation. Prehabilitation aims to optimize a patient before they undergo a major surgery. These programs combine exercise training, with nutritional optimization and psychological support. Together, these contribute to improve their muscle mass, tolerance to exercise, and nutritional status. The current study will assess whether an individualized and structured prehabilitation program combining supervised exercise training, nutritional optimization and psychological support will benefit patients with cirrhosis awaiting liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Diagnosis of cirrhosis, based on a combination of clinical, laboratory, imaging, or histology
* Active on the liver transplant waiting list of the MUHC

Exclusion Criteria:

* Biological Model for End Stage Liver Disease >20
* Hepatic decompensation within the last month
* High risk varices not on primary or secondary prevention
* Recurrent large volume paracentesis
* Persistent hepatic encephalopathy
* Platelets <20,000/µL, or hemoglobin <80g/L
* Altered hemodynamics
* Significant heart disease
* Awaiting combined organ transplantation
* Awaiting repeat liver transplantation
* Condition limiting mobilization and/or exercise, or recurrent falls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | 12 months
  Proportion of participants that adhere to the intervention protocol

SECONDARY OUTCOMES:
Safety of the intervention | 24 weeks
  Incidence of intervention-related adverse events
Impact of exercise program on frailty | At end of week-4, week-14, and week-24
  Interval change in liver frailty index, where a higher value indicates a higher degree of frailty
Impact of nutritional program on nutritional status | At end of week-4, week 14, and week-24
  Interval change in Royal Free Hospital Global Assessment status, where participants are classified as well nourished, moderately malnourished, or severely malnourished
Impact of psychological program on health-related quality of life | At end of week-4, week 14, and week-24
  Interval change in the Chronic Liver Disease Questionnaire (CLDQ) score where lower values indicate worse health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Amine Benmassaoud, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benmassaoud A, Gillis C, Geraci O, Martel M, Awasthi R, Barkun J, Chen T, Edgar L, Sebastiani G, Carli F, Bessissow A. Prehabilitation in patients with cirrhosis awaiting liver transplantation: protocol of a feasibility study. BMJ Open. 2024 Jun 25;14(6):e081362. doi: 10.1136/bmjopen-2023-081362. PMID 38925705